| <b>Document Type:</b> | Statistical Analysis Plan |
|---|---|
| Official Title: | A single arm, open-label, multicenter Phase 2 study of regorafenib in participants who have been treated in a previous Bayer-sponsored regorafenib study (monotherapy or combination treatment) that has reached the primary completion endpoint or the main data analysis, or has been stopped prematurely. |
| NCT Number: | NCT03890731 |
| <b>Document Date:</b> | 23 JUN 2023 |



BAY 73-4506 / 20328

## Title page

A single arm, open-label, multicenter Phase 2 study of regorafenib in participants who have been treated in a previous Bayer-sponsored regorafenib study (monotherapy or combination treatment) that has reached the primary completion endpoint or the main data analysis, or has been stopped prematurely.

## [Regorafenib rollover study]

Bayer study drug BAY 73-4506 / Regorafenib

**Study purpose:** Enable patients from the feeder studies to continue treatment

Clinical study II Date: 23 JUN 2023

phase:

**Study No.:** 20328 **Version:** 2.0

Author: PPD ,

ClinStat GmbH

### Confidential

The information provided in this document is strictly confidential and is intended solely for the guidance of the clinical investigation. Reproduction or disclosure of this document, whether in part or in full, to parties not associated with the clinical investigation or its use for any other purpose without the prior written consent of the sponsor is not permitted.

Throughout this document, symbols indicating proprietary names (®, TM) are not displayed. Hence, the appearance of product names without these symbols does not imply that these names are not protected.

This Statistical Analysis Plan is produced on a word-processing system and bears no signatures.

The approval of the Statistical Analysis Plan is documented in a separate Signature Document.

# BAY 73-4506 / 20328

# **Table of Contents**

| Titl | le page | 1 |
|---|---|---|
| Tal | able of Contents | |
| Abl | breviationsbreviations | 2 |
| 1. | Introduction | |
| 2. | Study Objectives | |
| 3. | Study Design | |
| 4. | General Statistical Considerations | 3 |
| 4.1 | General Principles | |
| 4.2 | Handling of Dropouts | 3 |
| 4.3 | Handling of Missing Data | 3 |
| 4.4 | Interim Analyses and Data Monitoring | 4 |
| 4.5 | Data Rules | 4 |
| 4.6 | Blind Review | 4 |
| <b>5.</b> | Analysis Sets | 4 |
| 5.1 | Assignment of analysis sets | |
| 6. | Statistical Methodology | 4 |
| 6.1 | Population characteristics | |
| 6.2 | Concomitant medication | |
| 6.3 | Study drug exposure | 5 |
| 6.4 | Efficacy | 5 |
| 6.5 | Pharmacokinetics/pharmacodynamics | 5 |
| 6.6 | Safety | |
| 6.7 | Subgroup analysis | 5 |
| 7. | Document history and changes in the planned statistical analysis | 5 |
| 8. | References | 6 |

# **Abbreviations**

| Tibble viacions | |
|-----------------|-----------------------------------------------------------|
| AE | Adverse event |
| ATC | WHO Anatomical Therapeutic Chemical Classification system |
| CRF | Case Report Form |
| ICF | Informed Consent Form |
| MedDRA | Medical Dictionary for Regulatory Activities |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| TEAE | Treatment-emergent adverse event |
| TESAE | Treatment-emergent serious adverse event |

### 1. Introduction

The primary purpose of the study is to enable participants, currently receiving regorafenib in a Bayer sponsored clinical trial, to continue treatment after their respective study has been completed. A completed study is defined as one that has reached the primary completion endpoint for main data analysis, or has been stopped prematurely, and the respective data have been cleaned. Participants will be able to continue treatment until the treating physician feels the participant is no longer benefiting from treatment.


### 2. **Study Objectives**

## Primary

The primary purpose of the program is to enable participants, currently receiving regorafenib in a Bayer sponsored clinical trial and assessed by the principal investigator (PI) to be benefitting, to continue regorafenib treatment after their respective study has met its primary completion date, or main data analysis, or has been stopped prematurely.

### Secondary

Documentation of safety and tolerability

### **3**. **Study Design**

This is an open label, single arm study.

#### 4. **General Statistical Considerations**

### 4.1 **General Principles**

The statistical evaluation will be performed by using the software package SAS release 9.2 or higher (SAS Institute Inc., Cary, NC, USA). All variables will be analyzed by descriptive statistical methods. The number of data available and missing data, mean, standard deviation, minimum, quartiles, median, and maximum will be calculated for metric data. Frequency tables will be generated for categorical data.

Due to the low number of expected patients no subgroup analyses are planned.

### 4.2 **Handling of Dropouts**

All data available will be analyzed.

### 4.3 **Handling of Missing Data**

All missing or partial data will be presented in the subject data listing as they are recorded on the Case Report Form (CRF).

The number of subjects who prematurely discontinue the study and study treatment for any reason, as well as the reasons for premature discontinuation of study and study treatment, will be reported.

## 4.4 Interim Analyses and Data Monitoring

Not applicable

### 4.5 Data Rules

In general all analyses will be performed for the safety set. It is anticipated that the analysis sets will not differ. Otherwise valuable data wich is not available in the safety set will also be analysed. See section 5 for definition of the analysis sets.

## 4.6 Blind Review

As this is an open label study, no unblinding is necessary. Patients will be assigned to the relevant analysis sets based on the rules described in section 5 for the analysis sets. This will be discussed and documented in the Blind Review Meeting.

## 5. Analysis Sets

For purposes of statistical analysis, the following analysis sets are defined:

| Analysis set | Description |
|---|---|
| Enrolled | All participants who signed the ICF |
| Safety | All participants who take at least 1 dose of regorafenib within this rollover study. |

## 5.1 Assignment of analysis sets

Assignment of the subjects to the analysis sets will be made based on the available treatment information (i.e. if there is a record indicating that regorafenib was taken, a patient will be assigned to the safety set).

## 6. Statistical Methodology

The main objective of the study is to ensure continuation of treatment for eligible patients and only safety data are collected. Beyond summary statistics, no statistical analysis is planned.

## 6.1 Population characteristics

If applicable, the number of subjects in each analysis set will be presented.

Due to the low number of patients expected in this study, no further summary statistics will be produced. Demographic data will be provided by means of a summary table and individual subject data listingsdisplaying the collected demographic informations as per CRF for all patients enrolled.

## 6.2 Concomitant medication

Concomitant medication will be analyzed in the safety set.

The frequency of concomitant medications will be summarized by 1<sup>st</sup> and 3<sup>rd</sup> level ATC class. This table will be repeated for concomitant anti-cancer therapy, if applicable.

### BAY 73-4506 / 20328

### 6.3 Study drug exposure

Study drug exposure will be analyzed in the safety set.

Treatment duration will be summarized as well as the number of applications and modifications of the study drug.


#### 6.4 **Efficacy**

Not applicable

### 6.5 Pharmacokinetics/pharmacodynamics

Not applicable

### 6.6 Safety

All analyses will be conducted in the safety set.

AEs will be coded using the latest version of MedDRA during the study. A treatmentemergent adverse event (TEAE) is defined as an AE that increase in severity or that is newly developed after the first study intervention.

If the onset date of an AE is missing/incomplete, it is assumed to have occurred after the first study intervention (i.e., a TEAE) except if the partial onset date or stop date indicates differently.

An overview over all patients experiencing AEs will be given. The total number of patients experiencing TEAEs will be presented and tabulated by SOC and PT and CTCAE grade.

The following categories will be presented:

- TEAEs
- Drug-related TEAEs
- TEAEs leading to discontinuation of study drug
- Treatment-emergent serious adverse events (TESAEs
- Drug-related TESAEs
- TESAEs leading to discontinuation of study drug

All deaths, TESAEs, TEAEs leading to discontinuation and pregnancies will be presented in subject listings, if applicable.

### 6.7 Subgroup analysis

Due to the low sample size no subgroup analysis will be conducted.

### 7. Document history and changes in the planned statistical analysis

This is the second version of the SAP. In comparison to the first version analysis were updated du to the small number of patients entering the study.

Reference Number: RD-SOP-1119

Supplement Version: 10

# **Statistical Analysis Plan**


# BAY 73-4506 / 20328

# 8. References

Final study protocol of study 20328, version 2.0, dated 20 NOV 2018 Final CRF of study 20328, dated 11 NOV 2020 SAP version 1, dated 28 MAR 2019